CLINICAL TRIAL: NCT02053454
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Single Ascending Dose, Safety, Tolerability and Pharmacokinetics Study of ALN-TTR02 in Japanese Healthy Volunteers
Brief Title: A Study of the Safety, Tolerability and Pharmacokinetics of ALN-TTR02 in Japanese Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALN-TTR02-005
Record Dates: First submitted 2014-01-24; First posted 2014-02-03 (Estimated); Last update posted 2015-05-25 (Estimated); Status verified 2015-05

CONDITIONS: Transthyretin (TTR)-Mediated Amyloidosis
Keywords: RNAi therapeutic
MeSH Terms: interventions — patisiran

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- patisiran (ALN-TTR02) (Active Comparator)
  Interventions: Drug: patisiran (ALN-TTR02)
- Sterile Normal Saline (0.9% NaCl) (Active Comparator)
  Interventions: Drug: Sterile Normal Saline (0.9% NaCl)

INTERVENTIONS:
Drug: patisiran (ALN-TTR02) — Ascending doses administered by intravenous (IV) infusion
  Arms: patisiran (ALN-TTR02)
Drug: Sterile Normal Saline (0.9% NaCl) — Calculated volume to match active comparator
  Arms: Sterile Normal Saline (0.9% NaCl)

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and pharmacokinetics (PK) of patisiran (ALN-TTR02) in Japanese subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy Japanese adult males and females aged 20 to 65 years, inclusive (The subject was born in Japan and has lived outside of Japan for <10 years, and subject's biological parents and grandparents are fully Japanese and were born in Japan);
* Subjects who are healthy as determined by clinical assessments;
* Females subjects must be of non-childbearing potential;
* Males with partners of child-bearing potential, must agree to use appropriate contraception.

Exclusion Criteria:

* Subjects with a history of serious mental illness;
* Subjects who have a clinically relevant medical or surgical history;
* Subjects with a positive screen for alcohol or drugs of abuse;
* Subjects with safety laboratory test results deemed clinically significant;
* Subjects with known hepatitis B surface antigen (HBsAg), hepatitis B virus (HBV), hepatitis C virus (HCV) or human immunodeficiency virus (HIV) infection;
* Subjects who have received an investigational agent within the 3 months prior to study entry.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-01; Primary Completion 2014-03 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects experiencing adverse events (AEs), serious adverse events (SAEs) and study drug discontinuation | Up to 28 days

SECONDARY OUTCOMES:
Pharmacodynamics (PD) of ALN-TTR02 (serum concentrations of Transthyretin, Vitamin A, and Retinol Binding Protein) | Up to 90 days
Observed maximum concentration (Cmax) of ALN-TTR02 | Up to 90 days
Time of observed maximum concentration (tmax) of ALN-TTR02 | Up to 90 days
Area under the plasma concentration versus time curve (AUC) of ALN-TTR02 | Up to 90 days
Terminal elimination half-life (t1/2) of ALN-TTR02 | Up to 90 days
Systemic clearance (CL) of ALN-TTR02 | Up to 90 days
Volume of distribution (V) of ALN-TTR02 | Up to 90 days
Renal clearance (CLR) of ALN-TTR02 | Up to 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Jared Gollob, MD, Study Director — Alnylam Pharmaceuticals
Locations (1):
- Clinical Site, London, United Kingdom